CLINICAL TRIAL: NCT04286100
Title: Comparison of Image Quality Generated by Contrast Specific Echocardiogram and Left Ventricular Opacification (LVO) Imaging Settings in Patients Enrolled in Luminity 422 Study
Brief Title: Contrast Specific Echocardiogram Versus Left Ventricular Opacification (LVO) Imaging Settings
Acronym: ELVIS
Status: Active, not recruiting | Type: Observational
Sponsor: London North West Healthcare NHS Trust (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: CRC/2019/002
Record Dates: First submitted 2020-01-13; First posted 2020-02-26 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Contrast Echocardiography Imaging
Keywords: Coronary artery disease; Myocardial contrast echocardiography; Left ventricle opacification
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study compares "contrast specific imaging setting" images with "left ventricular opacification (LVO)" images taken on the same group of patients at different points in time, to see if one is more effective at assessing the function of the heart.

DETAILED DESCRIPTION:
Ultrasound testing of the heart using a "dye" or contrast is often used to get clear pictures of the heart in many heart conditions. When this test is done when the heart is working hard, such as when exercising, this is called contrast stress echocardiography.

Current guidelines recommend the method called "contrast specific imaging setting," as the best way of looking at the main pumping part of the heart. However, it is not known if it provides better pictures when compared to a different method called "left ventricular opacification (LVO)."

This study will compare pictures in patients who have had tests done using both ways of looking at the heart and will compare; LVO; enhanced and unenhanced LVEBD; LVO imaging with contrast specific imaging Wall Motion Classification and LVO to contrast specific imaging Left Ventricular Ejection Fraction (LVEF). The comparison will be done by a group of experts in cardiac ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. Participants enrolled in the Luminity 422 study that also have complete data with contrast specific imaging obtained within a 60 day window.
2. Participants who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.

Exclusion Criteria:

1. Unwilling / unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From the 120 patients enrolled in the Luminity 422 clinical trial a cohort of participants underwent independent contrast specific imaging as part of their clinical management, during the time of recruitment for the trial. The contrast specific imaging data of these patients will be used.
  Sixty participants from the total of one hundred twenty patients that participated in the Luminity 422 clinical trial are planned to be enrolled in the study. They will have undergone further clinical echocardiographic assessment for other clinical reasons using the recommended contrast specific imaging setting by the same vendor.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To determine whether the technique left ventricular opacification (LVO) imaging provide better quality images than current best practice "contrast specific imaging setting," in patients routinely referred for a transthoracic echocardiogram. | 8 months

SECONDARY OUTCOMES:
To determine whether the technique LVO imaging provide better quality images than the current best practice for comparison of segmental LVEBD between images obtained by LVO imaging (intermediate MI) and contrast specific imaging (low MI). | 8 months
To determine whether the technique LVO imaging provide better quality images than the current best practice for comparison of wall motion classification between images obtained by LVO imaging (intermediate MI) and contrast specific imaging (low MI). | 8 months
To determine whether the technique LVO imaging provide better quality images than the current best practice for comparison of LVEF assessment between images obtained by LVO imaging (intermediate MI) and contrast specific imaging (low MI). | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Roxy Senior, Principal Investigator — LNWH Trust
Locations (1):
- Northwick Park Hospital, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No